CLINICAL TRIAL: NCT04136639
Title: The Anticariogenic Effect of Miswak (Silvadora Persica) and Grape Seed Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hala Ahmed Abdel Moneim, Principle Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC17-082
Record Dates: First submitted 2019-10-19; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Proanthocyanidins; Fluorides; Sodium Fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Miswak (Experimental): Miswak sticks used twice daily, every 12 hours, for three months.
  Interventions: Other: Miswak
- Grape Seed Extract (Experimental): Grape seed extract 6.5% mouthwash used twice daily, every 12 hours, for three months.
  Interventions: Other: Grape Seed Extract Mouthwash
- Fluoride Mouthwash (Active Comparator): 0.05% fluoride mouthwash used twice daily, every 12 hours, for three months.
  Interventions: Other: fluoride

INTERVENTIONS:
Other: Miswak — sticks
  Other Names: silvadora persica
  Arms: Miswak
Other: Grape Seed Extract Mouthwash — Mouthwash
  Other Names: 95% proanthocyanidins
  Arms: Grape Seed Extract
Other: fluoride — mouthwash
  Other Names: 0.05% sodium fluoride
  Arms: Fluoride Mouthwash

SUMMARY:
Prevention of dental caries has taken a great importance in the last decade. The use of herbal and natural products became mandatory to avoid the side effects of commercially available medications. Aim of the study; the aim was to investigate the anti-cariogenic effect of miswak and grape seed extract (GSE).

DETAILED DESCRIPTION:
Patients used Miswak sticks, grape seed extract mouth wash and fluoride mouthwash twice daily for three month. Saliva samples were collected at base line and after one month and three month. Assessment of bacterial count and saliva buffering capacity were performed at base line and after one and three month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high caries risk
* Males or females
* Medically free patients
* Patients approving to participate in the study

Exclusion Criteria:

* Patients who were on antibiotic therapy or corticosteroid therapy for 30 days before the examination
* Patients had history of professional cleaning in the last 15 days
* Patients with exposed pulp
* Evidence of parafunctional habits
* Patients with developmental dental anomalies
* Patients undergoing or will start orthodontic treatment
* Patients with removable prosthesis
* Periapical Abscess or Fistula

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
quantitative measure of the change in salivary streptococcus mutans Count from baseline to one month and three months. | Baseline, one month, three months.
  the patients used the treatments twice daily for three months. unstimulated saliva samples were collected from the patients at baseline,after one month and after three months. Every time samples were incubated with Mitiis Salivaris with Bacitricin and 20% sucrose for streptococcus mutans count.

SECONDARY OUTCOMES:
quantitative measure of the change in saliva buffering capacity from baseline to one month and three months. | baseline, one month , three months
  the patients used the treatments twice daily for three months. unstimulated saliva samples were collected from the patients at baseline, after one month and after three months. each time, saliva buffering capacity was measured using Hand Held pH meter and 0.1 mol/l hydrochloric acid that was titrated to the tested saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Niazy, Professor, Study Director — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No